CLINICAL TRIAL: NCT02967081
Title: Evaluation of Dentinal Fluid for the Presence of Matrix Metalloproteinase 9 (MMP-9) in Pulpal Inflammation
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: PB_2016-02043
Record Dates: First submitted 2016-11-11; First posted 2016-11-17 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Pulpitis
Keywords: Pulpitis; Biomarker; Diagnostic; Dentinal fluid
MeSH Terms: conditions — Pulpitis; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Pulp necrosis
  Interventions: Procedure: Collection of dentinal fluid using a cellulose membrane
- Pulpitis (painless): In this group the dentinal fluid will be sampled/collected twice: Firstly after the removal of the primary caries lesion. Subsequently the cavity will be temporized. Secondly, after removal of the temporary filling material (before final restoration).
  Interventions: Procedure: Collection of dentinal fluid using a cellulose membrane
- Irreversible pulpitis
  Interventions: Procedure: Collection of dentinal fluid using a cellulose membrane
- Normal pulp
  Interventions: Procedure: Collection of dentinal fluid using a cellulose membrane

INTERVENTIONS:
Procedure: Collection of dentinal fluid using a cellulose membrane — After removal of the caries lesion/filling a cellulose membrane (sterile paper point) will be applied with its blunt end to the dentin for 1 min to collect dentinal fluid.

SUMMARY:
The purpose of this study is to determine whether dentinal fluid (tooth fluid) of teeth with or without a painful inflammatory condition in their nerve (pulp) contain inflammatory marker.

DETAILED DESCRIPTION:
Objective:

The aim of the study is to use an improved sampling method for collection of MMP-9 to test the hypothesis that MMP-9 levels are significantly elevated in the dentinal fluid of symptomatic (painful) human permanent teeth compared to asymptomatic counterparts that need replacement of a filling, and pulp necrotic teeth. Moreover, the dynamics of MMP-9 expression after removal of the causative stimulus for pulpitis is to be investigated.

Outcome:

Measuring the total MMP-9 levels of dentinal fluid collected during dental treatment using a human MMP-9 fluorescent assay.

Measurements and procedures:

Patients attending the day service of the Center of Dental Medicine Zurich will be screened. Patients matching the inclusion criteria will be asked to participate in the study. Upon written informed consent, the affected tooth gets anesthetized, isolated with rubber dam and receives one of the following treatment procedures: caries removal and restoration, tooth filling replacement and restoration, or root canal treatment (because of irreversible pulpitis, or pulp necrosis). After caries removal, removal of the defect tooth filling, or during access cavity preparation, a cellulose membrane (paper point) will be applied with its blunt end to the dentin for 1 min to collect dentinal fluid. The cellulose membrane will be stored until the laboratory analysis. Depending on the individual treatment plan of the patient, the tooth will subsequently receive root canal treatment, its final restoration, or a temporization with glass-ionomer cement for coverage of the dentinal wound and reinforcement of the remaining tooth structure. Final restoration of a tooth with composite, a partial crowns, or full-coverage crown can be technically demanding, time consuming, and frequently involves multiple patient visits. Teeth that receive root canal treatment, or the final restoration are sampled once. When a patient with a temporized tooth returns for the final restoration, the sampling procedure (appliance of a cellulose membrane to the dentin for 1 min and storage for further analyses) will be repeated. Any further treatment will be continued without further impairments. The investigation does not alter the treatment plan of any patient (either participating in one, or two sampling procedures, or in the study at all).

Number of participants:

Based on a previously performed study (Zehnder et al., 2011), which used a similar experimental set-up and had 31 participants (2 groups), it is aimed to recruit 60 participants for the current study.

Comparators:

MMP-9 levels in dentinal fluid sampled from teeth with painful (irreversible) pulpitis will be compared to MMP-9 levels of teeth without clinical signs and symptoms. Moreover, the MMP-9 levels of teeth showing an painless pulpitis (teeth affected by a caries lesion) will be compared to a repeated sample of the same tooth collected after removal of the caries lesion.

Statistical analysis:

MMP-9 contents in the clinical samples will be determined against a standard curve (4-parameter logistic curve fit) obtained from the recombinant pro-MMP-9 standard dilution series. Values between groups will be compared by using Mann-Whitney U test, with the alpha-type error set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

Adult patients who attend the University of Zurich, Center of Dental Medicine, Clinic of Preventive Dentistry, Periodontology and Cariology that are in need for

* Treatment of pain related to pulpal inflammation
* Caries therapy
* Root canal treatment of a pulp-necrotic tooth
* Replacement of an defect/fractured filling

Exclusion Criteria:

* Children or adolescents (≤18 y)
* Patients who do not agree to participate in the study
* Patients with general diseases of inflammatory nature (such as diabetes, Crohn's disease, etc), or diseases affecting the immune-system (immuno-suppression, multiple morbidities, etc.)
* Women with known pregnancy
* Patients not fluent in German or English language
* Patients who had antibiotic or NSAID intake during the last 14 days
* Patients who refuse to be examined radiographically.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 y) who attend the University of Zurich, Center of Dental Medicine, Clinic of Preventive Dentistry, Periodontology and Cariology for dental treatment.
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2016-10; Primary Completion 2017-10-17 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
Total matrix metalloproteinase 9 (MMP-9) level in dentinal fluid | Immediately

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zurich, Center of Dental Medicine, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zehnder M, Wegehaupt FJ, Attin T. A first study on the usefulness of matrix metalloproteinase 9 from dentinal fluid to indicate pulp inflammation. J Endod. 2011 Jan;37(1):17-20. doi: 10.1016/j.joen.2010.10.003. PMID 21146069